CLINICAL TRIAL: NCT00275509
Title: Open Label Randomized Study of Thymoglobulin Versus Daclizumab Induction Therapies for the Reduction of Acute Rejection in Live Donor Kidney Transplant Recipients With a Positive Crossmatch
Brief Title: Induction Therapy Study in Live Donor Kidney Transplant Recipients With a Positive Crossmatch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00078055
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Kidney Failure, Chronic
Keywords: kidney; transplantation; positive crossmatch; antibody mediated rejection; rejection; induction; therapy; trial
MeSH Terms: conditions — Kidney Failure, Chronic; Rejection, Psychology | interventions — thymoglobulin; Daclizumab; Plasmapheresis; Mycophenolic Acid; Tacrolimus; Dexamethasone; Prednisone; cytomegalovirus-specific hyperimmune globulin

ARMS (2):
- Thymoglobulin (Experimental): Thymoglobulin was administered as 1.5 mg/kg prior to reperfusion followed by 6 post-operative doses on days 1 through 6.
  Interventions: Drug: Thymoglobulin; Other: Plasmapheresis; Drug: Mycophenolate mofetil; Drug: Tacrolimus; Drug: Dexamethasone; Drug: Prednisone; Drug: Cytogam
- Daclizumab (Experimental): Daclizumab was administered as 2 mg/kg prior to reperfusion followed by 1 mg/kg every other week for 8 weeks post-operatively (4 post-operative doses).
  Interventions: Drug: Daclizumab; Other: Plasmapheresis; Drug: Mycophenolate mofetil; Drug: Tacrolimus; Drug: Dexamethasone; Drug: Prednisone; Drug: Cytogam

INTERVENTIONS:
Drug: Thymoglobulin
  Arms: Thymoglobulin
Drug: Daclizumab
  Arms: Daclizumab
Other: Plasmapheresis — Following each plasmapheresis session, 100 mg/kg of Cytogam (CMVIg) (Cytogam, CSL Behring, King of Prussia, PA) was administered
Drug: Mycophenolate mofetil — 2 gm/day. Standard of care
Drug: Tacrolimus — To achieve serum level of 8-10 ng/ml.
Drug: Dexamethasone — 100 mg intra-operatively, and 25 mg every 6h post-operatively for six doses
Drug: Prednisone — Taper over three months to 5 mg daily
Drug: Cytogam — Following each plasmapheresis session, 100 mg/kg of Cytogam (CMVIg) (Cytogam, CSL Behring, King of Prussia, PA) was administered

SUMMARY:
The purpose of this study is to determine whether the anti-T cell antibody, Thymoglobulin is a more effective induction medication than the anti-IL-2R inhibitor daclizumab, in kidney transplant recipients who have a positive crossmatch with their live donor.

DETAILED DESCRIPTION:
Kidney transplantation is widely recognized as the optimal therapy for the management of end-stage renal disease. Presently, the deceased donor kidney waiting list has expanded disproportionately with the number of transplant procedures that are performed in the United States. To further compound this problem, as many as 1/3 of the patients on this list are highly sensitized against a broad range of potential donors.

In order to address this problem, we developed an antibody depletion protocol that permits transplantation in patients who have a positive crossmatch with their live donor. The protocol consists of standard immunosuppressant therapy, plasmapheresis, and intravenous immunoglobulin infusion. We have successfully performed transplantation in over 100 such patients with low complication rates.

Because these patients have been exposed to their donor's human leukocyte antigen (HLA) they are at high risk for both acute cellular and acute antibody-mediated rejection. This intent of this prospective, randomized, open-label trial is to determine whether induction therapy (i.e. therapy given at the time of transplantation for prophylaxis) with Thymoglobulin is associated with a lower 6-month incidence of acute cellular and antibody-mediated rejection than with our standard therapy, daclizumab.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older)
* End-stage renal disease
* Identified to have positive lymphocytotoxic crossmatch or flow cytometric crossmatch with live donor

Exclusion Criteria:

* Deceased donor recipients
* Pregnancy
* Active infection
* History of cancer within the past two years (with the exception of non-melanomatous skin cancer)
* History of heparin induced thrombocytopenia
* Medical contraindications to transplant procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Montgomery, M.D., Ph.D., Principal Investigator — Johns Hopkins University , SOM; Christopher E Simpkins, M.D., Study Director — Johns Hopkins University, SOM
Locations (1):
- The Johns Hopkins University, School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Haas M, Sis B, Racusen LC, Solez K, Glotz D, Colvin RB, Castro MC, David DS, David-Neto E, Bagnasco SM, Cendales LC, Cornell LD, Demetris AJ, Drachenberg CB, Farver CF, Farris AB 3rd, Gibson IW, Kraus E, Liapis H, Loupy A, Nickeleit V, Randhawa P, Rodriguez ER, Rush D, Smith RN, Tan CD, Wallace WD, Mengel M; Banff meeting report writing committee. Banff 2013 meeting report: inclusion of c4d-negative antibody-mediated rejection and antibody-associated arterial lesions. Am J Transplant. 2014 Feb;14(2):272-83. doi: 10.1111/ajt.12590. PMID 24472190
- [Background] Solez K, Colvin RB, Racusen LC, Haas M, Sis B, Mengel M, Halloran PF, Baldwin W, Banfi G, Collins AB, Cosio F, David DS, Drachenberg C, Einecke G, Fogo AB, Gibson IW, Glotz D, Iskandar SS, Kraus E, Lerut E, Mannon RB, Mihatsch M, Nankivell BJ, Nickeleit V, Papadimitriou JC, Randhawa P, Regele H, Renaudin K, Roberts I, Seron D, Smith RN, Valente M. Banff 07 classification of renal allograft pathology: updates and future directions. Am J Transplant. 2008 Apr;8(4):753-60. doi: 10.1111/j.1600-6143.2008.02159.x. Epub 2008 Feb 19. PMID 18294345

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 207 participant were assessed for eligibility. Excluded (n=151) Not meeting inclusion criteria (n=115) Declined to participate (n=2) Did not reach transplant prior to end of study (n=34). A total of 56 were randomized.
Period: Overall Study
Arm/Group | Thymoglobulin | Daclizumab
Started | 30 | 26
Completed | 30 | 25
Not Completed | 0 | 1
Not completed — graft thrombosis, post-operative day #8 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Tymoglobulin: Thymoglobulin was administered as 1.5 mg/kg prior to reperfusion followed by 6 post-operative doses on days 1 through 6
- Total: Total of all reporting groups
Arm/Group | Tymoglobulin | Daclizumab | Total
Number analyzed (Participants) | 30 | 26 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (10.6) | 46.5 (15.4) | 47.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 11 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 30 | 26 | 56

OUTCOME MEASURES:

1. Primary Outcome: 6-month Acute Cellular-mediated Rejection Rate (CMR)
Description: Per 2007 international Banff Classification Criteria, CMR 1A was diagnosed on biopsies displaying significant interstitial infiltration (>25% of parenchyma affected, i2 or i3) and foci of moderate tubulitis (t2). CMR IB was diagnosed in cases with significant interstitial infiltration (>25% of parenchyma affected, i2 or i3) and foci of severe tubulitis (t3). CMR IIA were cases with mild-to-moderate intimal arteritis (v1), while CMR IIB were those with severe intimal arteritis comprising >25% of the luminal area (v2). CMR III were those cases with transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic inflammation (v3).
Time Frame: Up to 6 months
Population: One patient in the Thymoglobulin arm died on post-operative day #8, prior to undergoing a biopsy. There were other deaths in the study however there were incidences of CMR, AMR or both prior to death.
Measure: Count of Participants; unit: Participants
Arm/Group | Tymoglobulin | Daclizumab
Number analyzed (Participants) | 29 | 26
Participants | 14 | 20

2. Primary Outcome: 6-month Acute Antibody-mediated Rejection Rate (AMR)
Description: A diagnosis of AMR was based on the 2013 international Banff Classification Criteria and is defined as the presence of circulating donor-specific antibody (DSA) and either: 1) peritubular capillary staining of C4d and at least one of the following: peritubular capillaritis (ptc) score>0, glomerulitis (g) score>0, acute thrombotic microangiopathy (TMA) in the absence of any other cause, or other features consistent with AMR (endothelial injury, fibrin thrombi, microinfarctions, interstitial hemorrhage), or 2) absence of capillary staining of C4d and the presence of ptc>0 and g>0 or ptc>0 or g>0 and acute TMA, in the absence of any other cause of TMA.
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tymoglobulin | Daclizumab
Number analyzed (Participants) | 29 | 26
Participants | 17 | 16

3. Primary Outcome: 6-month Cumulative Rejection Incidence (Either CMR, AMR or Both)
Description: Biopsy shows evidence of either AMR or CMR or evidence both.
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tymoglobulin | Daclizumab
Number analyzed (Participants) | 29 | 26
Participants | 21 | 23

ADVERSE EVENTS:
Time Frame: One year from date of transplant
Description: occasional assessment/testing
Arm/Group | Tymoglobulin | Daclizumab
All-Cause Mortality (participants affected / at risk) | 3/30 | 2/26
Serious Adverse Events (participants affected / at risk) | 6/30 | 9/26
Other Adverse Events (participants affected / at risk) | 19/30 | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tymoglobulin (N=30) | Daclizumab (N=26)
intra-thoracic vascular injury during placement of a central venous catheter (Surgical and medical procedures) | 1 (1) | 0 (0)
Allograft loss (Renal and urinary disorders) | 2 (2) | 4 (4)
Perforated gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cardiovascular disease (Cardiac disorders) | 1 (1) | 0 (0)
H1N1 flu (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus (RSV) Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Recurrent focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cytomegalovirus (CMV) (Infections and infestations) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Histoplasmosis (Infections and infestations) | 1 (1) | 3 (3)
Pancreatitis (General disorders) | 1 (1) | 0 (0)
Rejection (Product Issues) | 1 (2) | 0 (0)
Polyoma virus (BK) (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (UTI) (Infections and infestations) | 1 (1) | 1 (1)
delirium tremens seizure (General disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tymoglobulin (N=30) | Daclizumab (N=26)
Urinary Tract Infection (Infections and infestations) | 12 (17) | 9 (18)
Blood stream infection (Infections and infestations) | 1 (1) | 3 (3)
C-difficile infection (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Central line-associated bloodstream infection (CLABSI) (Infections and infestations) | 1 (1) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection of disc space (Infections and infestations) | 0 (0) | 1 (1)
Intra-abdominal infection (Infections and infestations) | 5 (6) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Polyoma virus (BK) (Infections and infestations) | 2 (2) | 1 (1)
Surgical site infection (Infections and infestations) | 3 (3) | 5 (6)
Upper respiratory infection (URI) (Infections and infestations) | 1 (4) | 2 (2)
Vancomycin-resistant enterococci (VRE) (Infections and infestations) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Rash (General disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Increase in creatinine (Renal and urinary disorders) | 1 (1) | 0 (0)
Bile infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes